CLINICAL TRIAL: NCT04258618
Title: CBT-I Targeting Co-morbid Insomnia in Patients Receiving RTMS for Treatment-Resistant Major Depressive Disorder
Brief Title: Cognitive Behavioral Therapy for Insomnia with RTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Drug Abuse Research Training Program (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00089725
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Depression; Insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I (Cognitive Behavioral Therapy for Insomnia) with TMS (Active Comparator)
  Interventions: Behavioral: CBT-I (Cognitive Behavioral Therapy for Insomnia) with rTMS
- rTMS (repetitive Transcranial Magnetic Stimulation) (Other): Subjects will be getting Transcranial Magnetic Stimulation as part of their standard of care.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Behavioral: CBT-I (Cognitive Behavioral Therapy for Insomnia) with rTMS — Cognitive Behavioral Therapy for insomnia (CBT-I) with rTMS (repetitive Transcranial Magnetic Stimulation) will be performed as part of this study by the PI. This includes weekly, one hour sessions addressing sleep for 6 weeks.
  Arms: CBT-I (Cognitive Behavioral Therapy for Insomnia) with TMS
Device: Repetitive Transcranial Magnetic Stimulation — Participants in this study will be undergoing repetitive transcranial magnetic stimulation (rTMS) for major depressive disorder as part of their clinical treatment. This involves magnetic stimulation with specific settings to a specific region of the brain to help treat depression. Treatment time ranges, but is around 30 minutes per session and occurs 5 days a week for 6 weeks.
  Arms: rTMS (repetitive Transcranial Magnetic Stimulation)

SUMMARY:
Depression and insomnia occur together in a substantial number of patients. Transcranial magnetic stimulation (TMS) is an effective treatment for depression, but does not help insomnia symptoms in depressed patients. A form of cognitive behavioral therapy (CBT) has been developed that specifically helps with insomnia (CBT-I). The study team will give CBT-I to patients who are being treated with TMS for depression, who also have insomnia, to determine if it helps insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years old
* Patients starting rTMS treatment for MDD
* Co-morbid insomnia as determined by meeting the following criteria: (a) Requiring more than 30 minutes to fall asleep at the beginning of the night or more than 30 minutes of time awake after initially falling asleep for at least 3 nights per week for at least 3 months - - An insomnia severity index score of 15 or more
* Manifested sleep disturbances or associated daytime symptoms causing significant distress or impairment in social, occupational or other areas of functioning
* Reliable access to a computer with internet access.

Exclusion Criteria:

* Obligation to an irregular sleep schedule that prevents the adoption of intervention strategies such as shift workers
* Participants who have received or are receiving CBT-I targeting insomnia in the past, or those who have initiated a new sedative medication, or sedating antidepressant within 2-weeks preceding enrollment
* Comorbid psychiatric disorders, including bipolar disorder, psychotic disorders or depression with psychotic features
* Presence of another untreated sleep disorder such as obstructive sleep apne
* Pregnancy
* Active substance use disorder within the past 3 months
* Use of medications that reduce the seizure threshold including Buproprion, stimulants or augmenting thyroid medications (for those without history of hypothyroid)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Reported Unanticipated Adverse Events | Baseline through post intervention (6 weeks)
  Tolerability of CBT-I with TMS determined by patient reported adverse event as assessed by red cap form
Percentage of patients completing CBT-I program | Determined post intervention (6 weeks)
  Feasibility of implementation of CBT-I as assessed by completion percentage of patients enrolled.

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale | Baseline and post intervention (6 weeks)
  Assessing pre and post TMS treatment changes of ESS in TMS + CBT-I group vs no CBT-I group. The scale is scored 0-24 assessing degree of sleepiness. Cutoff scores are as follows: 0-7:It is unlikely that you are abnormally sleepy. 8-9:You have an average amount of daytime sleepiness; 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention;16-24:You are excessively sleepy and should consider seeking medical attention. This scale is often used clinically for obstructive sleep apnea, but can be useful to assess daytime impact of insomnia.
Change in Insomnia Severity Index Scale | Baseline through post intervention (6 weeks)
  Assessing pre and post TMS treatment changes of ISI in TMS + CBT-I group vs no CBT-I group. This scale is scored 0-28 and is used to assess severity of insomnia with cutoff scores as follows: 0-7 = No clinically significant insomnia; 8-14 = Subthreshold insomnia;15-21 = Clinical insomnia (moderate severity); 22-28 = Clinical insomnia (severe).
Change in Patient Health Questionnaire - 9 | Baseline through post intervention (6 weeks)
  Assessing pre and post TMS treatment changes of PHQ-9 in TMS + CBT-I group vs no CBT-I group. This scale is used to assess depression severity. Cutoff scores are as follows: 0-4: Minimal or none; 5-9: Mild; 10-14: Moderate; 15-19: Moderately severe; 20-27: Severe.
Change in Pittsburgh Sleep Quality Index | Baseline and post intervention (6 weeks)
  Assessing pre and post TMS treatment changes of PSQI in TMS + CBT-I group vs no CBT-I group. This scale is a 9-item questionnaire assessing sleep quality. The score is determined by adding up 7 components, with a score of 5 or greater being considered poor sleep.
Change in Hamilton Rating Scale for Depression 17 | Baseline and post intervention (6 weeks)
  Assessing pre and post TMS treatment changes of HRSD 17 in TMS + CBT-I group vs no CBT-I group. This is a 17- item scale assessing severity of depression symptoms and is scored out of 58 (8 questions scored out of 5 and 9 questions scored out of 2), with 0-7 considered normal and > 20 considered at least moderate severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Norred, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norred MA, Haselden LC, Sahlem GL, Wilkerson AK, Short EB, McTeague LM, George MS. TMS and CBT-I for comorbid depression and insomnia. Exploring feasibility and tolerability of transcranial magnetic stimulation (TMS) and cognitive behavioral therapy for insomnia (CBT-I) for comorbid major depressive disorder and insomnia during the COVID-19 pandemic. Brain Stimul. 2021 Nov-Dec;14(6):1508-1510. doi: 10.1016/j.brs.2021.09.007. Epub 2021 Sep 23. No abstract available. PMID 34563744